CLINICAL TRIAL: NCT02167295
Title: Biobehavioral and Cultural Determinants of Betel Quid Chewing, Dependence, and Withdrawal in Taiwan
Acronym: BCDBQCDWT
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Cheng-Chieh Lin, Attending physician, China Medical University Hospital
Other Study IDs: DMR101-IRB1-258(CR-2)
Record Dates: First submitted 2013-02-26; First posted 2014-06-19 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Smoking; Betel Nut
Keywords: betel nut; dependence; withdraw; deprivation test
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The urine of participants for self-report questionnaire study will be retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Focus group: The focus groups will consist of 6 to 8 persons each (N = 32). The focus group discussions will last for about 60 to 90 minutes. The discussion topics will be based on previous literature and experience and will include reasons for betel quid chewing or for quitting, pros and cons of betel quid chewing, barriers to and facilitators of abstinence, health beliefs and experiences about betel quid chewing and other issues.
- In-depth interviews.: We will conduct 15 one-to-one interviews, each lasts for about 45 to 60 minutes. Participants will be interviewed by a trained interviewer using a structured interview. The interview will be designed to collect information on socio-demographic background, current and/or former betel quid use, other substance use (smoking and/or alcohol consumption), as well as other variables including usage parameters, psychosocial and environmental influences on betel quid chewing, barriers to and interest in quitting, and knowledge of adverse effects on health.
- Self-report questionnaire: This study is expected to enroll 30 participants who have smoking and betel nut chewing behaviors.Participants will complete 4 separate visits to CMUH, during which they will complete the same self-report questionnaire designed to measure withdrawal symptoms relating to betel quid chewing. To better measure betel quid withdrawal symptoms and to distinguish the 6 symptoms from those of smoking withdrawal, Participants will be required to attend one visit regular cigarette smoking and betel nut chewing behavior without restriction (as control), one visit after 12 hours of overnight betel quid deprivation (no cigarette deprivation), one visit after 12 hours of overnight cigarette deprivation (no betel quid deprivation), and one visit after 12 hours of both overnight betel quid and cigarette deprivation.

SUMMARY:
Cancer of the oral cavity is one of the fastest growing cancers among men in Taiwan. Previous research has established a strong link between betel quid chewing, a common practice among Taiwanese men, and oral cancer. However, despite the strong association, no attempt has been made to develop behavioral measures to facilitate betel quid cessation. This application extends upon existing collaboration between MD Anderson and China Medical University Hospital (CMUH) and seeks to characterize betel quid chewers and their withdrawal symptoms, in order to address an urgent cancer epidemiology issue in Taiwan.

DETAILED DESCRIPTION:
Cancer of the oral cavity is one of the fastest growing cancers among men in Taiwan. Previous research has established a strong link between betel quid chewing, a common practice among Taiwanese men, and oral cancer. However, despite the strong association, no attempt has been made to develop behavioral measures to facilitate betel quid cessation. This application extends upon existing collaboration between MD Anderson and China Medical University Hospital (CMUH) and seeks to characterize betel quid chewers and their withdrawal symptoms, in order to address an urgent cancer epidemiology issue in Taiwan. In a two phase study, we will use a qualitative approach (guided focus group and interviews), followed by assessment of betel quid withdrawal in current chewers: 1) 47 participants will be invited to participate in a qualitative study that includes focus group and in-depth structured interviews that examine the social and cultural context that surrounds continued use and cessation of betel quid consumption, 2) 30 male and female healthy individuals who currently both chew betel quid and smoke cigarettes will be invited to attend 4 separate sessions at CMUH and complete a self-report questionnaire specifically designed to measure betel quid withdrawal symptoms, and the relationship between betel quid chewing and cigarette smoking withdrawal. This application represents the first step in the development of a multi-phase, multidisciplinary betel quid chewing research program. This program will enhance our understanding of the cultural and bio-behavioral aspects of betel quid chewing. Furthermore, it will lead to translational research projects that link behavioral findings to clinical treatments, and the eventual creation of a large scale, population-based prevention and education program.

ELIGIBILITY:
Inclusion Criteria:

* Smoking and betel nut chewing habit and at least 20 years old to 65 years old and healthy people.

Exclusion Criteria:

* 1. Less than 20 years old or greater than 65 years.
* 2. No smoking and betel nut chewing habit.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. 47 participants will be invited to participate in a qualitative study that includes focus group and in-depth structured interviews that examine the social and cultural context that surrounds continued use and cessation of betel quid consumption.
  2. 30 male and female healthy individuals who currently both chew betel quid and smoke cigarettes will be invited to attend 3 separate sessions at CMUH and complete a self-report questionnaire specifically designed to measure betel quid withdrawal symptoms, and the relationship between betel quid chewing and cigarette smoking withdrawal. This application represents the first step in the development of a multi-phase, multidisciplinary betel quid chewing research program.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Predictive validity of a self-reported measure of areca nut dependency scale. | up to 28days

SECONDARY OUTCOMES:
Develop a self-report questionnaire that examines betel quid withdrawal | focus group each lasts for about 60 to 90 minutes and one-to-one interviews each lasts for about 45 to 60 minutes.
  To know reasons for betel quid chewing or for quitting, pros and cons of betel quid chewing, barriers to and facilitators of abstinence, health beliefs and experiences about betel quid chewing and other issues.And then, we propose to develop a self-report questionnaire that examines betel quid withdrawal among Taiwanese chewers who are also current cigarette smokers.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan